CLINICAL TRIAL: NCT00165191
Title: A Phase II Study of Doxorubicin, Cisplatin, and 5-Fluorouracil in Patients With Advanced Adenocarcinoma of the Stomach or Esophagus
Brief Title: Doxorubicin, Cisplatin, 5-Fluorouracil in Patients With Advanced Adenocarcinoma of the Stomach or Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-048
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Adenocarcinoma of Stomach; Adenocarcinoma of GE Junction; Adenocarcinoma of Esophagus
Keywords: doxorubicin; cisplatin; 5-fluorouracil; stomach cancer; esophagus cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms; Esophageal Neoplasms | interventions — Doxorubicin; Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: Doxorubicin
Drug: Cisplatin
Drug: 5-fluorouracil

SUMMARY:
The purpose of this study is to collect information on the anti-tumor activity of the combination doxorubicin, cisplatin, and 5-fluorouracil when given to patients with advanced esophageal or gastric adenocarcinoma. We will also be collecting information about the side effects and safety of this combination.

DETAILED DESCRIPTION:
* Patients will receive cisplatin and doxorubicin intravenously once every 3 weeks. In addition to cisplatin and doxorubicin, patients will receive 5-fluorouracil intravenously as a continuous infusion for the duration of the study. In order to do this, patients will receive an infusion pump that can be carried with them. Treatment cycles will be repeated every 21 days for a maximum of 8 cycles.
* Prior to enrollment in this study and while the patient is receiving the therapy, routine blood tests and x-ryas (including chest x-rays and CT scans) will be performed to check the body's response to the treatment. Blood tests will be checked once a week and chest x-rays and CT scans will be checked every 6 weeks.
* Patients with progressive disease or intolerable side effects will be removed from the study. Patients with stable disease or tumor response will continue therapy for a maximum of 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Measurable, locally unresectable or metastatic adenocarcinoma of the stomach, GE junction or esophagus
* No more than one prior chemotherapy regimen
* ECOG performance status of < or equal to 2
* Life expectancy > 12 weeks
* ANC > 1,500/mm3
* Hemoglobin > 9.0 gm/dl
* Platelets > 100,000/mm3
* SGOT < 3 x ULN
* Total bilirubin < 2.0 mg/dl
* Creatinine < 1.5 mg/dl

Exclusion Criteria:

* Prior cisplatin or doxorubicin as neoadjuvant or adjuvant therapy with in 1 year of study entry
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Myocardial infarction in the past 6 months
* Major surgery in the past 2 weeks
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women
* Concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History or clinical evidence of congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 1998-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To determine the activity of doxorubicin, cisplatin and continuous infusion of 5-fluorouracil in patients with measurable, locally unresectable or metastatic adenocarcinoma of the stomach, GE junction, or esophagus.

SECONDARY OUTCOMES:
Assess the safety of doxorubicin, cisplatin and 5-fluorouracil when given in combination to treat this patient population
evaluate the survival of this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts